CLINICAL TRIAL: NCT06721481
Title: Radiofrequency Electromagnetic Fields and Pregnancy : Exposure Specificities and Evolution: the RFM - Expo Study
Brief Title: Radiofrequency Electromagnetic Fields and Pregnancy : Exposure Specificities and Evolution
Acronym: RFM - Expo
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Swiss Tropical and Public Health Institute (Switzerland) (Unknown); University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/923
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Radiofrequencies Exposure; Pregnancy; Real Life Study
Keywords: radiofrequencies; exposure science; exposure meter; 5G

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women who attend their first prenatal consultation at the maternity ward of the University hospital of Besançon

SUMMARY:
The purpose of this study is to investigate the specific features of radiofrequencies (RF) exposure (including 5G) in pregnant women, its evolution during pregnancy and the quantitative contribution of the various RF emission sources to which they are exposed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years of age;
* Subject not opposed to participating in the study;
* Patient performing the three screening ultrasounds recommended by the French National Authority for Health (HAS) at the Universitary hospital of Besançon during her pregnancy (independently or in addition to on-site clinical pregnancy monitoring); Affiliation with a French social security scheme or beneficiary of such a scheme; Living within the Universitary hospital of Besançon maternity catchment area, to cover the full range of geographical exposure, including both highly urbanized and more rural areas;

Exclusion Criteria:

* Opposition of the subject to participate in the study;
* Discontinuation of pregnancy ultrasound follow-up at Besançon University Hospital, in particular due to relocation;
* Women under court protection, guardianship, curatorship or protective supervision.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1,500 pregnant women having their first prenatal ultrasound visit at the maternity ward of the Besançon University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assessing the exposure of pregnant women to radiofrequencies | 3 days
  Women have to wear a personal portable exposure meter during 3 days.

SECONDARY OUTCOMES:
Quantifying the evolution of this exposure during pregnancy | 3 periods of 3 days
  The measurement is repeted for each trimester of pregnancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birks LE, Struchen B, Eeftens M, van Wel L, Huss A, Gajsek P, Kheifets L, Gallastegi M, Dalmau-Bueno A, Estarlich M, Fernandez MF, Meder IK, Ferrero A, Jimenez-Zabala A, Torrent M, Vrijkotte TGM, Cardis E, Olsen J, Valic B, Vermeulen R, Vrijheid M, Roosli M, Guxens M. Spatial and temporal variability of personal environmental exposure to radio frequency electromagnetic fields in children in Europe. Environ Int. 2018 Aug;117:204-214. doi: 10.1016/j.envint.2018.04.026. Epub 2018 May 10. PMID 29754001